CLINICAL TRIAL: NCT04993391
Title: A Dose-escalation, Dose-extension and Efficacy-extension, Phase I/II Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Profile and Preliminary Efficacy of AP-L1898 Capsule for the Treatment of the Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer
Brief Title: AP-L1898 Capsule in Patients With Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Suzhou Junjing BioSciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS111-001-I
Record Dates: First submitted 2021-06-10; First posted 2021-08-06 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-08

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 40mg dose. (Experimental): The subjects will receive a single dose at first in this stage, and be observed for 7 days subsequently, if tolerated, the subjects will enter the multi-dose study on oral AP-L1898 once per day for consecutive 21 days. The DLT observational per
  Interventions: Drug: JS111(AP-L1898 Capsules)
- 80mg dose. (Experimental): The subjects will receive a single dose at first in this stage, and be observed for 7 days subsequently, if tolerated, the subjects will enter the multi-dose study on oral AP-L1898 once per day for consecutive 21 days. The DLT observational per
  Interventions: Drug: JS111(AP-L1898 Capsules)
- 160mg dose. (Experimental): The subjects will receive a single dose at first in this stage, and be observed for 7 days subsequently, if tolerated, the subjects will enter the multi-dose study on oral AP-L1898 once per day for consecutive 21 days. The DLT observational pe
  Interventions: Drug: JS111(AP-L1898 Capsules)
- 240mg dose. (Experimental): The subjects will receive a single dose at first in this stage, and be observed for 7 days subsequently, if tolerated, the subjects will enter the multi-dose study on oral AP-L1898 once per day for consecutive 21 days. The DLT observational pe
  Interventions: Drug: JS111(AP-L1898 Capsules)
- 320mg dose. (Experimental): The subjects will receive a single dose at first in this stage, and be observed for 7 days subsequently, if tolerated, the subjects will enter the multi-dose study on oral AP-L1898 once per day for consecutive 21 days. The DLT observational pe
  Interventions: Drug: JS111(AP-L1898 Capsules)

INTERVENTIONS:
Drug: JS111(AP-L1898 Capsules) — 40 mg, QD
  Arms: 40mg dose.
Drug: JS111(AP-L1898 Capsules) — 80 mg, QD
  Arms: 80mg dose.
Drug: JS111(AP-L1898 Capsules) — 160 mg, QD
  Arms: 160mg dose.
Drug: JS111(AP-L1898 Capsules) — 240 mg, QD
  Arms: 240mg dose.
Drug: JS111(AP-L1898 Capsules) — 320 mg, QD
  Arms: 320mg dose.

SUMMARY:
This is a phase I/II, open-label, first-in-human clinical study designed to evaluate the safety, tolerability, PK profile and efficacy of JS111 for patients with Non-small cell lung cance. This study is divided into 3 periods: dose escalation stage, dose extension stage, and efficacy extension stage.

ELIGIBILITY:
"Inclusion criteria:

1. Age≥18 years, male or female;
2. Patients with histologically or cytologically confirmed locally advanced (stage IIIB/IIIC) or metastatic (stage IV) NSCLC that can not undergo radical chemoradiotherapy;
3. Dose-escalation and dose-extension periods: failure of standard of care or intolerance of standard of care, having received at least one or more systemic therapeutic regimens for locally advanced or metastatic disease;
4. There is clear evidence showing carrying EGFR exon 20 insertion and other rare EGFR mutations (only applicable for dose-extension and efficacy-extension periods). The test method can use: ARMS method for tissue or cell specimen (need to be tested in national certified laboratory), NGS method for tissue or blood specimen (need to be tested in CLIA or CAP certified laboratory). Note: enrollment of patients does not need to be confirmed by central laboratory;
5. At least one measurable lesion meeting RECIST v1.1 definition, no history of puncture biopsy for the target lesion within the previous two weeks;
6. United States Eastern Cooperative Oncology Group (ECOG) Performance Status score 0~1;
7. Life expectancy >12 weeks;
8. Having adequate function of important organs at screening (requiring no blood transfusion, no use of hematopoietic stimulating factor or human albumin preparation within 14 days prior to screening):

   1. Absolute neutrophil count (ANC) ≥1.5x109/L;
   2. Platelets ≥100×109/L;
   3. Haemoglobin > 90 g/L;
   4. Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5×upper limit of normal (ULN) (for known liver metastasis, ≤ 5×ULN);
   5. Total bilirubin ≤1.5×ULN;
   6. Coagulation function INR≤1.5 ULN;
   7. Serum creatinine ≤ 1.5×ULN or creatinine clearance (Ccr, calculated using Cockcroft-Gault formula) ≥45 mL/min;
   8. Serum lipase and amylase ≤ 1.5 × ULN;
9. Serum pregnancy test must be confirmed as negative for women of childbearing potential within 7 days prior to enrollment, who agree upon use of effective contraceptive measures during use of the study drug and within 6 months after the last dose. Women of childbearing potential in this protocol is defined as sexually mature women: 1) no hysterectomy or bilateral ovariectomy, 2) uncontinuous natural menopause for 24 months (i.e., menses occurred at any time in the previous consecutive 24 months; fertility can not be excluded in case of amenorrhoea following cancer therapy). Male subjects whose partners are women of childbearing potential must agree to take effective contraceptive measures during the use of study drug and within 6 months after the last dose;
10. Being voluntary to participate in this study after sufficient informed consent and sign the informed consent form.

Exclusion criteria:

1. Use of any chemotherapeutic agen within 14 days prior to the first dose of AP-L1898; or the time from discontinuation of other investigational product to the use of anticancer drug less than 5 half-lives or 28 days, whichever is shorter;
2. EGFR exon 20 insertion cohort in efficacy-extension stage: once used the drugs targeting EGFR exon 20 insertion mutation (e.g., AZD9291, TAK-788, Poziotinib, CLN-081, JNJ-372, etc.); the patients previously receiving AZD9291 for treatment of EGFR sensitive mutation are allowed to be enrolled;
3. Ongoing use of CYP3A potent inhibitor or inducer, or discontinuation of potent inhibitor less than 5 half-lives of the drug, or discontinuation of potent inducer less than 5 half-lives of the drug or 14 days (whichever is longer) at the first dose of AP-L1898;
4. Not recovered from the adverse event induced by previous antitumor therapy at screening (recovered to ≤ grade 1) (except alopecia);
5. Having other malignant tumors within 5 years prior to the start of treatment or simultaneously (except radically treated non-melanoma without evidence on recurrence of disease, including skin basal cell carcinoma or squamous cell carcinoma, breast/cervical carcinoma in situ, superficial bladder cancer and other carcinomas in situ);
6. Presence of active gastrointestinal disease or other conditions that may obviously affect absorption, metabolism or excretion of drugs;
7. Patients who known to have received organ transplantation;
8. Major surgery performed within 28 days prior to the first dose. Small surgery permitted, e.g., minimally invasive biopsy;
9. Patents with carcinomatous meningitis, spinal cord compression at present;
10. At rested state, mean corrected QT interval QTc, using Fridericia's correction formula>450 ms in man or >470 ms in woman on electrocardiography (ECG) (repeated for three times). A variety of clinically significant abnormalities in cardiac rhythm, conduction or morphology of resting ECG, e.g., complete left bundle branch block, degree III heart block, degree II heart block, PR interval>250 ms. Any factors that may increase the risk of prolonged QTc interval or risk of arrhythmic events, e.g., heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in lineal relatives, or ongoing use of any drug known to prolong QT interval;
11. History of poorly controlled hypertension;
12. Previous history of the following diseases: interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis requiring steroid therapy, active interstitial lung disease with clinical evidence;
13. Patients with active brain metastasis, if the CNS metastasis is only limited to supratentorial area or cerebellum that has been adequately treated (surgery or radiotherapy) and radiologically stable for at least 4 weeks, and no corticosteroid is needed to control symptoms, the patients will be allowed to be enrolled;
14. In acute infection phase and requiring pharmacotherapy;
15. HBV DNA≥103 copies/mL or ≥200 IU/mL when the hepatitis B surface antigen is positive or hepatitis B core antibody is positive;
16. HCV-RNA > the upper limit of reference at the site when hepatitis C antibody is positive;
17. Human immunodeficiency virus (HIV) antibody positive;
18. Patient with a previous history of clear mental disorder and taking drugs for treatment;
19. Patient with a history of drug abuse or drug taking;
20. Pregnant or lactating women;
21. Presence of other factors that may possibly affect the study results, interfere with their participation in the entire study, including previous or current physical condition (e.g., ocular disease, including corneal ulcer, conjunctivitis, etc.), treatment or laboratory examination abnormality, unwillingness to comply with each procedure, restriction and requirement in the study, as considered by investigators.

A limited list of criteria for selection of participants in the clinical study, provided in terms of inclusion and exclusion criteria and suitable for assisting potential participants in identifying clinical studies of interest. Use a bulleted list for each criterion below the headers ""Inclusion Criteria"" and ""Exclusion Criteria"". (Limit: 15,000 characters.)"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2021-07-13 (Actual); Primary Completion 2024-06-18 (Estimated); Study Completion 2024-08-18 (Estimated)

PRIMARY OUTCOMES:
Safety assessed by the adverse event | up to 3 years
  The AEs summary will be provided.
Safety assessed by the serious adverse event | up to 3 years
  The SAEs summary will be provided.
Safety assessed by the physical examinatin | up to 3 years
  The abnormal physical examinatin summary will be provided.
Safety assessed by the ECOG score | up to 3 years
  The worsening ECOG score summary will be provided.
Safety assessed by the ophthalmic examination | up to 3 years
  The ophthalmic examination summary will be provided.
ORR | up to 3 years
  The ORR summary will be calculated.

SECONDARY OUTCOMES:
Cmax | 0up to 3 years
  observed maximum plasma concentration of AP-L1898
Tmax | up to 3 years
  time ro reach maximum plasam concentration of AP-L1898
AUC 0-t | up to 3 years
  Area under the concentration versus time curve from time 0 to the last measurable concentration (AUC 0-t)
t1/2 | up to 3 years
  Elimination half life time
CL/F | up to 3 years
  apparent clearance (CL/F)
Vd/F | up to 3 years
  Apparent volume of distribution (Vd/F)
DoR | up to 3 years
  the time from the first evaluation of CR or PR to the first evaluation of PD or death for any reason. For the subjects who have no progression but survive persistently after meeting the response criteria, the duration of response will be censored on the date of the last evaluable tumor evaluation or the last follow-up of progression of disease.
OS | up to 3 years
  Kaplan-Meimer method will be used to plot survival curve, while the median survival will be calculated.
DCR | up to 3 years
  the proportion of subjects with CR, PR or SD as the best response in accordance with RECIST1.1.
Plasma drug concentration after administration of study drug | up to 3 years
  The actual date and time of collection of each PK sample (24h system, accurate to minute) will be recorded in the study. Except an accurate record of the actual time point for collection of PK sample, the administration also needs to be recorded to evaluate PK data. The plasma concentrations of AP-L1898 and its metabolites will be determined using validated LC-MS/MS method.

CONTACTS AND LOCATIONS:
Locations (37):
- China (37):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Chinese People's Liberation Army Army Characteristic Medical Center, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Sun Yat-sen Memorial Hospital ], Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Cancer Hospital Chinese Academy of Medical Sciences，Shenzhen center, Shenzhen, Guangdong
  - Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong
  - Liuzhou People's Hospital, Liuchow, Guangxi
  - Harbin Medical University Cancer Hospital, Haerbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - North Jiangsu People's Hospital, Yangzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Neimenggu
  - Shandong Cancer Hospital, Jinan, Shandong
  - Weifang People's Hospital, Weifang, Shandong
  - Shanghai Oriental Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Hangzhou Cancer Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital , Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
  - Hunan Cancer Hospital, Changsha
  - Zhejiang Cancer Hospital, Hangzhou
  - Shanghai Pulmonary Hospital, Shanghai